CLINICAL TRIAL: NCT00959413
Title: Assessment of HIV-1-Related Oral Mucosal Disease and Use of Saliva in Measuring HIV-1 Viral Load
Brief Title: Assessing HIV-Related Oral Mucosal Disease and Using Saliva to Measure Viral Load
Status: Completed | Type: Observational
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG A5254; 1U01AI068636 (NIH)
Record Dates: First submitted 2009-08-12; First posted 2009-08-14 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples of saliva and blood will be kept
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A: Participants who have a CD4 count of 200 cells/mm3 or less and a viral load greater than 1,000 copies/ml
- B: Participants who have a CD4 count of 200 cells/mm3 or less and a viral load of 1,000 copies/ml or less
- C: Participants will have a CD4 count that is greater than 200 cells/mm3 and a viral load that is greater than 1,000 copies/ml
- D: Participants will have a CD4 count that is greater than 200 cells/mm3 and a viral load that is 1,000 copies/ml or less

SUMMARY:
The mouth may play an important part in monitoring HIV progression. Mucosal lesions of the mouth are often the first sign of infection and their development in already diagnosed individuals indicates disease progression. In addition, saliva may provide a non-invasive way to track viral load. The purpose of this study is to establish standardized practices for examining the mouth and identifying oral mucosal lesions as well as to establish a correlation of viral load with HIV particles found in saliva.

DETAILED DESCRIPTION:
The oral cavity has been found to play an important role in monitoring the progression of HIV infection. The occurrence of specific lesions, mainly oral candidiasis and hairy leukoplakia, is strongly associated with a low CD4 cell count and a higher plasma viral load. Furthermore, even though the prevalence of specific oral lesions like candidiasis, hairy leukoplakia, and Kaposi sarcoma (KS) has been found to be lower among patients on highly active antiretroviral therapy (HAART), other oral lesions such as warts have been found to be more prevalent in this population. In addition, saliva has been shown to harbor viral particles, antibodies, and cytokines, and may represent an easily and noninvasively collected specimen for various diagnostic assays, including early diagnosis of HIV. The purpose of this study is to establish a set of standardized practices for examining and diagnosing oral mucosal lesions and to establish a correlation between the amount of HIV found in the saliva with viral load.

Participants in this study will attend only one screening visit and study visit and will be assigned to one of four groups based on viral load and CD4 count. Group A will consist of participants who have a CD4 count of 200 cells/mm3 or less and a viral load greater than 1000 copies/ml. Group B will be made up of participants who have a CD4 count of 200 cells/mm3 or less and a viral load of 1000 copies/ml or less. Group C participants will have a CD4 count that is greater than 200 cells/mm3 and a viral load that is greater than 1000 copies/ml. Participants making up Group D will have a CD4 count that is greater than 200 cells/mm3 and a viral load that is 1000 copies/ml or less.

All participants will have a medical history taken and blood collected as well as performing a throat wash collection and whole saliva collection. In addition, two oral exams will be performed at the study visit.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, as documented by any rapid test or licensed ELISA test kit and confirmed by Western blot, HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA
* CD4+ cell count obtained ≤ 60 days prior to study entry
* Plasma HIV-1 RNA levels obtained ≤ 60 days prior to study entry
* If receiving ART, participants must be on same ART regimen for at least 12 weeks immediately prior to study entry
* If study participants are not currently on an ART regimen, they must have not discontinued ART therapy within 30 days prior to study entry
* Ability and willingness of study participant or legal guardian/representative to provide informed consent

Exclusion Criteria:

* History of head and/or neck radiation secondary to malignancy
* History of any HIV-1 therapeutic related vaccines
* Use of any systemic anti-fungal in the 90 days prior to entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected individuals
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Presumptive clinical diagnoses of oral mucosal diseases | At study visit
HIV-1 viral load in throat wash. | At study visit
HIV-1 viral load in plasma | At study visit
Candida CFU level as measured in CFU/mL of throat wash solution. | At study visit

SECONDARY OUTCOMES:
Prevalence of HIV-1 related oral mucosal lesions | At study visit
KSHV DNA viral load in throat wash | At study visit
CMV DNA load in throat wash | At study visit
Oral candidal genotypes | At study visit
Antifungal resistance as measured by MIC | At study visit
HSV-1 DNA viral load in throat wash | At study visit
EBV DNA viral load in throat wash | At study visit

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Aberg, MD, Study Chair — NYU Langone Health; Caroline Shiboski, DDS, MPH, PhD, Study Chair — Department of Orofacial Sciences, University of California, San Francisco
Locations (6):
- United States (5):
  - Ucsf Aids Crs (801), San Francisco, California
  - The Ponce de Leon Ctr. CRS (5802), Atlanta, Georgia
  - NY Univ. HIV/AIDS CRS (401), New York, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Case CRS (2501), Cleveland, Ohio
- Les Centres GHESKIO CRS (30022), Bicentenaire, Port-au-Prince, Haiti